CLINICAL TRIAL: NCT05261659
Title: Using Sleep and Dreaming to Treat Social Anxiety
Brief Title: Targeted Memory Reactivation During REM Sleep in Patients With Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Lampros Perogamvros, Senior Clinical Fellow, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-01335
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Social Anxiety Disorder; Sleep
MeSH Terms: conditions — Phobia, Social | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMR group (Experimental): Patients will receive a sound while they receive a positive feedback for their performance of exposure therapy (ET). They will also receive the sound during REM sleep.
  Interventions: Behavioral: Exposure Therapy and Targeted memory reactivation during REM sleep
- Control group (Active Comparator): Patients will not receive a sound while they receive a positive feedback for their performance of exposure therapy (ET). They will receive the same sound as the experimental group during REM sleep under the same conditions.
  Interventions: Behavioral: Exposure Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy and Targeted memory reactivation during REM sleep — Emerging evidence shows that REM sleep plays a causal role in extinction learning, emotion regulation and consolidation of emotionally positive memories. By using targeted memory reactivation (TMR), a known method where a sound is associated with a waking experience (i.e., positive feedback in this study) and strengthening it during REM sleep, the investigators aim to accelerate the remission of social anxiety disorder.
  Arms: TMR group
Behavioral: Exposure Therapy — These patients will receive the classic treatment of Exposure Therapy (ET) for social anxiety disorder without any association with a sound.
  Arms: Control group

SUMMARY:
With this study, the investigators aim to use sleep and dreaming in order to enhance exposure therapy for social anxiety disorder (SAD), by pairing the positive feedback phase of exposure (public talk) to an auditory stimulus during wake (associated sound) and subsequently applying this stimulus during sleep (targeted memory reactivation, TMR). Exposure therapy sessions will take place in a virtual reality (VR) environment, while physiological measures during the preparation phase of public talk such as heart rate variability (HRV), skin conductance response (SCR) and subjective level of anxiety (SUDS) will be used in order to assess treatment efficiency across the sessions. Patients with SAD according to DSM-5 criteria will be included.

The main hypothesis of this study is that participants who are presented with the associated sound during sleep (TMR group) will have reduced intensity of social anxiety compared to participants with no such association (control group), after both a full night's sleep with auditory stimulation during REM sleep in the laboratory, and after 1 week of stimulation during REM sleep at home. In addition, it is expected that fear-related dreams may correlate with anxiety levels during wakefulness after 1 week of stimulation at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients with social anxiety disorder (according to DSM-5 criteria and Liebowitz Social Anxiety Scale > 65)
* aged between 16 and 40 yo
* no current treatment for SAD (cognitive-behavioral therapy, medications)

Exclusion Criteria:

* mood disorder, psychosis,other anxiety disorder or other mental disorders according to DSM-5 criteria
* sleep disorder (e.g.,insomnia disorder, obstructive sleep apnea syndrome, restless legs syndrome) according to DSM-5 criteria
* use of psychiatric medication
* current treatment for SAD (cognitive-behavioral therapy, medications)
* neurological disease

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Root mean square of the successive [R-R intervals] differences | 1 day
  The RMSSD is used to estimate the vagally mediated changes in heart rate variability.
Root mean square of the successive [R-R intervals] differences | 1 week
  The RMSSD is used to estimate the vagally mediated changes in heart rate variability.
Subjective Units of Distress Scale | 1 day
  Validated rating of subjective distress on a scale of 0 to 10 (higher values reflect a worse outcome)
Subjective Units of Distress Scale | 1 week
  Validated rating of subjective distress on a scale of 0 to 10 (higher values reflect a worse outcome)

SECONDARY OUTCOMES:
Non-specific skin conductance responses | 1 day
  The skin conductance response measures sympathetic nervous system activation.
Non-specific skin conductance responses | 1 week
  The skin conductance response measures sympathetic nervous system activation.
Change of fear in dreams (average of fear during the second week with stimulations minus the first week without stimulations) | 1 week
  Use of a dream diary where the emotion of fear is graded in a dichotomous way (presence/absence).

OTHER OUTCOMES:
Liebowitz Social Anxiety Scale | 3 months
  Validated self-report measure used to assess degree of social anxiety on a scale of 0 to 144 (higher values reflect a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sleep Medicine, University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No